CLINICAL TRIAL: NCT00505388
Title: A Follow-up Programme for Patients Using Symbicort SMART in Normal Clinical Practice
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Other Study IDs: D5890C00018; EuDract 2006-005677-22
Record Dates: First submitted 2007-07-17; First posted 2007-07-23 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2010-04

CONDITIONS: Bronchial Asthma
Keywords: asthma; bronchial; Symbicort
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This patient follow-up programme was designed to describe the extent of Symbicort use in patients prescribed Symbicort as maintenance and reliever therapy in routine clinical practice in comparison with the already documented use of Symbicort as maintenance and reliever therapy in clinical therapies

ELIGIBILITY:
Inclusion Criteria:

* Asthma patients prescribed Symbicort as maintenance and reliever therapy, according to the label, before inclusion in this programme
* signed and dated informed consent(ICF)
* for patients under-age, signed and dated ICF form from both the patient and the patient's parent/legal guardian is required

Exclusion Criteria:

* Involvement in the planning and conduct of the programme (applies to both AstraZeneca staff or staff at the investigational site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients continued with their treatment (Symbicort SMART) after enrolment. Enrolment throug IVRS/IWRS, no randomisation. Primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 5137 (Actual)
Dates: Start 2007-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Andersson, MD, Study Director — AstraZeneca; Bjorn Stallberg, MD, Principal Investigator — Trosa Vardcentral
Locations (695):
- Belgium (220):
  - Research Site, Aarschot
  - Research Site, Achel
  - Research Site, Alleur
  - Research Site, Alsemberg
  - Research Site, Amay
  - Research Site, Angleur
  - Research Site, Ans
  - Research Site, Antheit (= Wanze)
  - Research Site, Antwerp
  - Research Site, Assenede
  - Research Site, Ath
  - Research Site, Aywaille
  - Research Site, Baal
  - Research Site, Begijnendijk
  - Research Site, Bellaire (beyne-heusay)
  - Research Site, Bellegem
  - Research Site, Belsele (sint-niklaas)
  - Research Site, Beringen
  - Research Site, Bertrix
  - Research Site, Betekom
  - Research Site, Beverst
  - Research Site, Beyne-Heusay
  - Research Site, Bilzen
  - Research Site, Binche
  - Research Site, Boechout
  - Research Site, Borgerhout
  - Research Site, Bornem
  - Research Site, Borsbeke
  - Research Site, Braine-l'Alleud
  - Research Site, Braine-le-Comte
  - Research Site, Brasschaat
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Brussels (anderlecht)
  - Research Site, Brussels (ganshoren)
  - Research Site, Brussels (ixelles)
  - Research Site, Brussels (laeken)
  - Research Site, Brussels (molenbeek-st-jean)
  - Research Site, Brussels (schaerbeek)
  - Research Site, Brussels (uccle)
  - Research Site, Brussels (watermaal-bosvoorde)
  - Research Site, Brussels (woluwe-st-pierre)
  - Research Site, Brustem
  - Research Site, Buggenhout
  - Research Site, Champion
  - Research Site, Chênée
  - Research Site, Couillet
  - Research Site, De Pinte
  - Research Site, Deinze
  - Research Site, Dendermonde
  - Research Site, Deurne (antwerpen)
  - Research Site, Diegem
  - Research Site, Diepenbeek
  - Research Site, Diksmuide
  - Research Site, Dottignies
  - Research Site, Dour
  - Research Site, Dranouter
  - Research Site, Duffel
  - Research Site, Dworp
  - Research Site, Eisden
  - Research Site, Ekeren
  - Research Site, Ensival
  - Research Site, Ertvelde
  - Research Site, Evergem
  - Research Site, Écaussinnes-d'Enghien
  - Research Site, Écaussinnes-Lalaing
  - Research Site, Feluy
  - Research Site, Genappe
  - Research Site, Genk
  - Research Site, Genly
  - Research Site, Geraardsbergen
  - Research Site, Ghent
  - Research Site, Ghlin
  - Research Site, Godinne
  - Research Site, Gozée
  - Research Site, Grivegnée
  - Research Site, Haine-Saint-Pierre
  - Research Site, Halen
  - Research Site, Halle
  - Research Site, Ham-sur-Heure
  - Research Site, Hamme (o-vl)
  - Research Site, Hamont
  - Research Site, Hasselt
  - Research Site, Havré
  - Research Site, Heist-op-den-Berg
  - Research Site, Heppen
  - Research Site, Herentals
  - Research Site, Herzele
  - Research Site, Heurne
  - Research Site, Heusden
  - Research Site, Hever
  - Research Site, Hoboken (antwerpen)
  - Research Site, Hoeselt
  - Research Site, Hooglede
  - Research Site, Houffalize
  - Research Site, Houthalen-Helchteren
  - Research Site, Hove
  - Research Site, Huldenberg
  - Research Site, Hulste
  - Research Site, Huy
  - Research Site, Jamioulx
  - Research Site, Keerbergen
  - Research Site, Kerkom
  - Research Site, Kessel
  - Research Site, Kobbegem
  - Research Site, Koolskamp
  - Research Site, Kortrijk
  - Research Site, Kraainem
  - Research Site, Kumtich
  - Research Site, Kuringen
  - Research Site, Landen
  - Research Site, Langdorp
  - Research Site, Leffinge
  - Research Site, Leopoldsburg
  - Research Site, Leut
  - Research Site, Libramont
  - Research Site, Lier
  - Research Site, Limbourg
  - Research Site, Linkebeek
  - Research Site, Lochristi
  - Research Site, Lommel
  - Research Site, Lustin
  - Research Site, Luttre
  - Research Site, Maasmechelen
  - Research Site, Maldegem
  - Research Site, Manage
  - Research Site, Marchovelette
  - Research Site, Mechelen
  - Research Site, Mechelen-aan-de-Maas
  - Research Site, Melsbroek
  - Research Site, Merelbeke
  - Research Site, Merksem (antwerpen)
  - Research Site, Meulebeke
  - Research Site, Middelkerke
  - Research Site, Moerkerke
  - Research Site, Mol
  - Research Site, Monceau-sur-Sambre
  - Research Site, Mons
  - Research Site, Mont-sur-Marchienne
  - Research Site, Moorsel
  - Research Site, Mortier
  - Research Site, Mouscron
  - Research Site, Munsterbilzen
  - Research Site, Natoye
  - Research Site, Neerpelt
  - Research Site, Nivelles
  - Research Site, Oostham
  - Research Site, Oostkamp
  - Research Site, Oostrozebeke
  - Research Site, Opgrimbie (maasmechelen)
  - Research Site, Opwijk
  - Research Site, Ostend
  - Research Site, Oudenaarde
  - Research Site, Overpelt
  - Research Site, Paal
  - Research Site, Perk
  - Research Site, Pittem
  - Research Site, Plancenoit
  - Research Site, Presles
  - Research Site, Puurs
  - Research Site, Quaregnon
  - Research Site, Ransart
  - Research Site, Rendeux
  - Research Site, Riemst
  - Research Site, Rijkevorsel
  - Research Site, Rijkhoven
  - Research Site, Rochefort
  - Research Site, Ronquières
  - Research Site, Ronse
  - Research Site, Rotem
  - Research Site, Rumst
  - Research Site, Saint-Médard
  - Research Site, Schuiferskapelle
  - Research Site, Sibret
  - Research Site, Sint-Baafs-Vijve
  - Research Site, Sint-Gillis-bij-Dendermonde
  - Research Site, Sint-Katherina-Lombeek
  - Research Site, Sint-Niklaas
  - Research Site, Sint-Truiden
  - Research Site, Spouwen (bilzen)
  - Research Site, Steendorp
  - Research Site, Steenokkerzeel
  - Research Site, Stekene
  - Research Site, Tavier
  - Research Site, Tessenderlo
  - Research Site, Theux
  - Research Site, Thuin
  - Research Site, Tielen
  - Research Site, Tielt
  - Research Site, Tienen
  - Research Site, Tienen (kumtich)
  - Research Site, Torhout
  - Research Site, Tournai
  - Research Site, Tremelo
  - Research Site, Trois-Ponts
  - Research Site, Uitkerke
  - Research Site, Verviers
  - Research Site, Veurne
  - Research Site, Villers-Poterie
  - Research Site, Vilvoorde
  - Research Site, Vorst
  - Research Site, Vrasene
  - Research Site, Vucht (maasmechelen)
  - Research Site, Waimes
  - Research Site, Waret-l'Évêque
  - Research Site, Weerde
  - Research Site, Welkenraedt
  - Research Site, Wespelaar
  - Research Site, Wezembeek-Oppem
  - Research Site, Wépion
  - Research Site, Wilsele
  - Research Site, Wingene
  - Research Site, Yvoir
  - Research Site, Zedelgem
  - Research Site, Zemst
  - Research Site, Zichen-Zussen-Bolder
  - Research Site, Zoersel
  - Research Site, Zolder
  - Research Site, Zomergem
  - Research Site, Zottegem
- Bulgaria (8):
  - Research Site, Blagoevgrad
  - Research Site, Kardzhali
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Razgrad
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Troyan Municipality
- Czechia (19):
  - Research Site, Brno
  - Research Site, Děčín
  - Research Site, Havířov
  - Research Site, Holice
  - Research Site, Hradec Králové
  - Research Site, Kladno
  - Research Site, Kolín
  - Research Site, Liberec
  - Research Site, Litoměřice
  - Research Site, Lovosice
  - Research Site, Most
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Prostějov
  - Research Site, Strakonice
  - Research Site, Teplice
  - Research Site, Ústí nad Labem
- Denmark (22):
  - Research Site, Aabenraa
  - Research Site, Aalborg
  - Research Site, Aså
  - Research Site, Birkerød
  - Research Site, Frederiksberg
  - Research Site, Frederikssund
  - Research Site, Kalundborg
  - Research Site, Kåstrup
  - Research Site, Kerteminde
  - Research Site, Kobenmhavn V
  - Research Site, Kolding
  - Research Site, Korsør
  - Research Site, København S
  - Research Site, Nakskov
  - Research Site, NYKoBING SaeLLAND
  - Research Site, Nærum
  - Research Site, Odense C
  - Research Site, Roskilde
  - Research Site, Rungsted
  - Research Site, Rødovre Municipality
  - Research Site, Solrød Strand
  - Research Site, Vordingborg
- Germany (160):
  - Research Site, Apolda
  - Research Site, Auerbach
  - Research Site, Augsburg
  - Research Site, Bad Berka
  - Research Site, Bad Salzuflen
  - Research Site, Bad Schwartau
  - Research Site, Bad Segeberg
  - Research Site, Bad Tölz
  - Research Site, Beelitz
  - Research Site, Bergisch Gladbach
  - Research Site, Bergkamen
  - Research Site, Berlin
  - Research Site, Beuel
  - Research Site, Blankenhain
  - Research Site, Bocholt
  - Research Site, Braunschweig
  - Research Site, Buchholz
  - Research Site, Burg
  - Research Site, Büchen
  - Research Site, Bützow
  - Research Site, Calbe/Saale
  - Research Site, Calvörde
  - Research Site, Cologne
  - Research Site, Cottbus
  - Research Site, Crinitz
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Düsseldorf
  - Research Site, Eisleben Lutherstadt
  - Research Site, Elsterwerda
  - Research Site, Engelskirchen-Runderoth
  - Research Site, Eppelborn
  - Research Site, Erfurt
  - Research Site, Essen
  - Research Site, Euskirchen
  - Research Site, Fehmarn / OT Burg
  - Research Site, Frankenthal
  - Research Site, Frankfurt
  - Research Site, Freiburg-Tiengen
  - Research Site, Freital
  - Research Site, Freudenberg
  - Research Site, Fuldatal
  - Research Site, Gars
  - Research Site, Gärtringen
  - Research Site, Geesthacht
  - Research Site, Genthin
  - Research Site, Gotha
  - Research Site, Grefrath
  - Research Site, Greven
  - Research Site, Grimma
  - Research Site, GroBenhain
  - Research Site, Gummersbach
  - Research Site, Hagen
  - Research Site, Haigerloch
  - Research Site, Haldensleben I
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hamm
  - Research Site, Hanau
  - Research Site, Hanover
  - Research Site, Hartha
  - Research Site, Heidelberg
  - Research Site, Heilbronn
  - Research Site, Hemmingen
  - Research Site, Hirschorn
  - Research Site, Homburg
  - Research Site, Horneburg
  - Research Site, Hückeswagen
  - Research Site, Hünxe
  - Research Site, Ibbenbueren
  - Research Site, Iffezheim
  - Research Site, Ilmenau
  - Research Site, Jühnde
  - Research Site, Karlsfeld
  - Research Site, Kassel
  - Research Site, Kelkheim
  - Research Site, Köthen
  - Research Site, Kronau
  - Research Site, Künzelsau
  - Research Site, Leipzig
  - Research Site, Leverkusen
  - Research Site, Liebenau
  - Research Site, Lienen
  - Research Site, Lippstadt
  - Research Site, Ludwigsburg
  - Research Site, Ludwigshafen
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, Mannheim
  - Research Site, Marburg
  - Research Site, Mendig
  - Research Site, Metzingen
  - Research Site, Mitteleschenbach
  - Research Site, Monheim
  - Research Site, Mülsen
  - Research Site, München
  - Research Site, Münster
  - Research Site, Nassau
  - Research Site, Netphen
  - Research Site, Neubrandenburg
  - Research Site, Neuruppin
  - Research Site, Neuss
  - Research Site, Neuwied
  - Research Site, Nordhausen
  - Research Site, Oberursel
  - Research Site, Oberwiesenthal
  - Research Site, Ochtrup
  - Research Site, Offenbach
  - Research Site, Osterburg
  - Research Site, Otterbach
  - Research Site, Ottweiler
  - Research Site, Paderborn
  - Research Site, Parey
  - Research Site, Pinneberg
  - Research Site, Plauen
  - Research Site, Potsdam
  - Research Site, Pretzien
  - Research Site, Pulsnitz
  - Research Site, Reinfeld
  - Research Site, Reinsdorf
  - Research Site, Remscheid
  - Research Site, Remscheid-Lennep
  - Research Site, Rheinberg
  - Research Site, Rüdersdorf
  - Research Site, Saalfeld
  - Research Site, Schleswig
  - Research Site, Schleusingen
  - Research Site, Schöneberg
  - Research Site, Schrobenhausen
  - Research Site, Schwaig
  - Research Site, Schweitzingen
  - Research Site, Siegen
  - Research Site, Sinsheim
  - Research Site, Solingen
  - Research Site, Sonneberg
  - Research Site, Sonneberg/Thuringen
  - Research Site, Sömmerda
  - Research Site, Spalt
  - Research Site, Speyer
  - Research Site, Suhl
  - Research Site, Sulzbach
  - Research Site, Sulzetal
  - Research Site, Teterow
  - Research Site, Thallwitz
  - Research Site, Trossingen
  - Research Site, Viersen
  - Research Site, VS-Villingen
  - Research Site, Wangen
  - Research Site, Wardenburg
  - Research Site, Warendorf
  - Research Site, Weilheim
  - Research Site, Weinheim
  - Research Site, Welbsleben
  - Research Site, Welver
  - Research Site, Wernigerode
  - Research Site, Wetter
  - Research Site, Willich
  - Research Site, Winsen
  - Research Site, Witten
  - Research Site, Zehdenick
- Greece (20):
  - Research Site, Agía Paraskeví
  - Research Site, Aigio
  - Research Site, Athens
  - Research Site, Cholargós
  - Research Site, Halkida
  - Research Site, Hraklion- Crete
  - Research Site, Irakleio
  - Research Site, Kalithèa
  - Research Site, Lamia
  - Research Site, Larissa
  - Research Site, Lávrio
  - Research Site, Marousi
  - Research Site, Metamorfosi
  - Research Site, Nafplion
  - Research Site, Néa Smýrni
  - Research Site, Pátrai
  - Research Site, Peristeri
  - Research Site, Ptolemaida
  - Research Site, Thessaloniki
  - Research Site, Zografou
- Hungary (17):
  - Research Site, Baja
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Dabas
  - Research Site, Debrecen
  - Research Site, Dunaújváros
  - Research Site, Gyula
  - Research Site, Kiskunhalas
  - Research Site, Komárom
  - Research Site, Komló
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Siófok
  - Research Site, Székesfehérvár
  - Research Site, Szombathely
  - Research Site, Tatabánya
  - Research Site, Zalaegerszeg
- Netherlands (84):
  - Research Site, 's-Gravenzande
  - Research Site, 's-Hertogenbosch
  - Research Site, Almelo
  - Research Site, Almere Stad
  - Research Site, Amersfoort
  - Research Site, Amstelveen
  - Research Site, Amsterdam
  - Research Site, Appingedam
  - Research Site, Arcen
  - Research Site, Beek en Donk
  - Research Site, Beilen
  - Research Site, Bergen op Zoom
  - Research Site, Berkel-Enschot
  - Research Site, Bunschoten
  - Research Site, Coevoerden
  - Research Site, Den Helder
  - Research Site, Denekamp
  - Research Site, Doetinchem
  - Research Site, Dordrecht
  - Research Site, Drachetn
  - Research Site, Duiven
  - Research Site, Edam
  - Research Site, Ede
  - Research Site, Eindhoven
  - Research Site, Enschede
  - Research Site, Ermelo
  - Research Site, Flushing
  - Research Site, Geleen
  - Research Site, Gouda
  - Research Site, Harderwijk
  - Research Site, Heel
  - Research Site, Heerlen
  - Research Site, Heeten
  - Research Site, Helmond
  - Research Site, Hengelo
  - Research Site, Hoogwoud
  - Research Site, Hulst
  - Research Site, Landgraaf
  - Research Site, Leeuwarden
  - Research Site, Lichtenvoorde
  - Research Site, Lieshout
  - Research Site, Losser
  - Research Site, Lunteren
  - Research Site, Maastricht
  - Research Site, Nijmegen
  - Research Site, Nijverdal
  - Research Site, Onstwedde
  - Research Site, Oud-Beijerland
  - Research Site, Oude Pekela
  - Research Site, Poortvliet
  - Research Site, Rijssen
  - Research Site, Rijswijk
  - Research Site, Rilland
  - Research Site, Roelofsarendsveen
  - Research Site, Roermond
  - Research Site, Rotterdam
  - Research Site, Ruinen
  - Research Site, Saint Willebrord
  - Research Site, Schiedam
  - Research Site, Sint-Michielsgestel
  - Research Site, Sittard
  - Research Site, Sneek
  - Research Site, Spijkenisse
  - Research Site, Swifterband
  - Research Site, The Hague
  - Research Site, Tilburg
  - Research Site, Tubbergen
  - Research Site, Ulft
  - Research Site, Urk
  - Research Site, Utrecht
  - Research Site, Vlaardingen
  - Research Site, Volendam
  - Research Site, Wassenaar
  - Research Site, Weert
  - Research Site, Westmaas
  - Research Site, Wildervank
  - Research Site, Winterswijk
  - Research Site, Woerden
  - Research Site, Wolvega
  - Research Site, Woudrinchem
  - Research Site, Zutphen
  - Research Site, Zwartmeer
  - Research Site, Zwijndrecht
  - Research Site, Zwolle
- Norway (33):
  - Research Site, Aksdal
  - Research Site, Arendal
  - Research Site, Avaldnes
  - Research Site, Årnes
  - Research Site, Bergen
  - Research Site, Elverum
  - Research Site, Fevik
  - Research Site, Fredrikstad
  - Research Site, Frogner
  - Research Site, Grimstad
  - Research Site, Hamar
  - Research Site, Haugesund
  - Research Site, Hovik
  - Research Site, Kirkeaer
  - Research Site, Kløfta
  - Research Site, Kolbjørnsvik
  - Research Site, Kongsberg
  - Research Site, Kristiansand
  - Research Site, Larvik
  - Research Site, Lierskogen
  - Research Site, Oslo
  - Research Site, Paradis
  - Research Site, Rådal
  - Research Site, Rykkin
  - Research Site, Skiptvet
  - Research Site, Spikkestad
  - Research Site, Srumsand
  - Research Site, Stavanger
  - Research Site, Strømmen
  - Research Site, Svelvik
  - Research Site, Tolvsrød
  - Research Site, Trondheim
  - Research Site, Ulset
- Portugal (17):
  - Research Site, Alfragide
  - Research Site, Almada
  - Research Site, Amadora
  - Research Site, Aveiro
  - Research Site, Barcarena
  - Research Site, Castelo Branco
  - Research Site, Charneca DA Caparica
  - Research Site, Coimbra
  - Research Site, Covilha
  - Research Site, Ermesinde
  - Research Site, Faro
  - Research Site, Lisbon
  - Research Site, Penafiel
  - Research Site, Porto
  - Research Site, Setúbal
  - Research Site, Torres Vedras
  - Research Site, Vila Nova de Gaia
- Sweden (43):
  - Research Site, Arlöv
  - Research Site, Arvidsjaur
  - Research Site, Avesta
  - Research Site, Åkersberga
  - Research Site, Åtvidaberg
  - Research Site, Borlänge
  - Research Site, Gothenburg
  - Research Site, Gullspång
  - Research Site, Helsingborg
  - Research Site, Höllviken
  - Research Site, Jarfalla
  - Research Site, Karlskrona
  - Research Site, Kil
  - Research Site, Kristianstad
  - Research Site, Kristinehamn
  - Research Site, Lidingö
  - Research Site, Lilla Edet
  - Research Site, Limhamn
  - Research Site, Linköping
  - Research Site, Ljusdal
  - Research Site, Ludvika
  - Research Site, Luleå
  - Research Site, Lyckeby
  - Research Site, Lycksele
  - Research Site, Malmo
  - Research Site, Partille
  - Research Site, Piteå
  - Research Site, Sollentuna
  - Research Site, Stenstorp
  - Research Site, Stockholm
  - Research Site, Storuman
  - Research Site, Svedala
  - Research Site, Trollhättan
  - Research Site, Trosa
  - Research Site, Tyreso
  - Research Site, Ullanger
  - Research Site, Upplands Vasby
  - Research Site, Vaxjo
  - Research Site, Vännäs
  - Research Site, Västerås
  - Research Site, Vellinge
  - Research Site, Vinslöv
  - Research Site, Ystad
- United Kingdom (52):
  - Research Site, Darlington, CO. Durham
  - Research Site, Hayle, Cornwall
  - Research Site, NR Penzance, Cornwall
  - Research Site, Penzance, Cornwall
  - Research Site, Keresley, Coventry
  - Research Site, Bexhill-on-Sea, EAST Sussex
  - Research Site, Glenrothes, Fife/scotland
  - Research Site, Bangor, Gwynedd
  - Research Site, Canterbury, KENT
  - Research Site, Dartford, KENT
  - Research Site, Motherwell, Lanarkshire
  - Research Site, Burbage, Leicester
  - Research Site, Wells-next-the-Sea, Norfolk
  - Research Site, Bangor, Northern Ireland
  - Research Site, CO Antrim, Northern Ireland
  - Research Site, Ecclesfield, Sheffield
  - Research Site, Barry, South Glamorgan
  - Research Site, Atherstone, Warwickshire
  - Research Site, Royal Leamington Spa, Warwks
  - Research Site, Walsall, WEST Midlands
  - Research Site, Crawley, WEST Sussex
  - Research Site, Chippenham, Wiltshire
  - Research Site, Corsham, Wiltshire
  - Research Site, Trowbridge, Wiltshire
  - Research Site, Westbury, Wiltshire
  - Research Site, Ashford
  - Research Site, Ashton-under-Lyne
  - Research Site, Ayrshire
  - Research Site, Bath
  - Research Site, Bathgate
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, Blantyre
  - Research Site, Bolton
  - Research Site, BURY Saint Edmonds
  - Research Site, Carrickfergus
  - Research Site, Coventry
  - Research Site, Doncaster
  - Research Site, Glasgow
  - Research Site, Hamilton
  - Research Site, Harrow
  - Research Site, Loughborough
  - Research Site, Minchinhampton
  - Research Site, NEW Stevenson
  - Research Site, Newcastle upon Tyne
  - Research Site, Peterborough
  - Research Site, Sheffield
  - Research Site, Stevenage
  - Research Site, Stockport
  - Research Site, Watford
  - Research Site, Welingborough

REFERENCES:
- [Derived] Stallberg B, Naya I, Ekelund J, Eckerwall G. Real-life use of budesonide/formoterol in clinical practice: a 12-month follow-up assessment in a multi-national study of asthma patients established on single-inhaler maintenance and reliever therapy. Int J Clin Pharmacol Ther. 2015 Jun;53(6):447-55. doi: 10.5414/CP202224. PMID 25907171